CLINICAL TRIAL: NCT03844152
Title: Investigating the Effect of Fermented Whey Concentrate on Gut Microbial Activity: Does Butyrate Matter?
Brief Title: RIGHTWHEY - Responders In Gut HealTh Markers Using Fermented WHEY
Acronym: RIGHTWHEY
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: University of Aberdeen (Other)
Collaborators: A. Vogel (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 808
Record Dates: First submitted 2019-01-29; First posted 2019-02-18 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Health, Subjective; Healthy; Microbial Colonization
Keywords: fermented whey; microbiota; gut health; butyrate
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Intervention Model Description: Stratified single arm study
Masking Description: The intervention will be provided in non-descript bottles. Fermented whey is mixed with sugar-free flavoured water to mask its taste from participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fermented whey concentrate (Experimental): Volunteers will receive the premixed water and fermented whey in weekly deliveries in 1.5L bottles and a drinking glass with a clear indication of the required 200ml volume. Participants will be asked to drink 200 ml of the supplemented water twice daily for the active intervention period.
  Interventions: Dietary Supplement: Fermented whey concentrate

INTERVENTIONS:
Dietary Supplement: Fermented whey concentrate — The investigated dietary supplement is a form of lacto-fermented whey concentrate (FWC), which has been deproteinised and then diluted (1/20) in sugar-free flavoured water to improve palatability. The main solute within the lacto-fermented whey is L-(+)-lactic acid (7%), produced through bacterial fermentation of the milk sugar lactose. The research team will provide non-descriptive bottles of drink to all volunteers. The flavour of the FWC will be masked by the flavoured water. In order to assess compliance and minimize an initial treatment effect, a 14 day run-in period during which only flavoured water is to be consumed will be completed by all volunteers. At the same time, this period will act as a wash-out, as volunteers will be asked to abstain from the use of any dietary supplements during this period and the rest of the study. The daily energy content of the FWC is 4kcal.
  Other Names: Molkosan

SUMMARY:
This 8-week intervention will investigate the effect of daily consumption of a fermented whey concentrate on the short-chain fatty acid profile of faeces in healthy individuals.

This study will help us understand if consumption of fermented foods rich in lactic acid have a beneficial effect on gut health.

DETAILED DESCRIPTION:
The 8-week dietary supplementation trial will investigate the action of exogenous lactic acid consumption on the activity (using short-chain fatty acid) and composition of the gut microbiota.

Participants will be stratified according to their baseline faecal butyrate levels. Therefore volunteers will be asked to provide two faecal samples one week apart. Based on the average absolute level of butyrate in the faecal samples, volunteers will be stratified into either low, moderate or high baseline butyrate levels (detailed in table 1 below). The levels for faecal butyrate for each group are set based on a meta-analysis of 9 human studies of healthy volunteers carried out at the Rowett Institute (n=116; LaBouyer et al, 2016, unpublished). Thresholds were derived from the boundaries of tertiles. Therefore, the moderate butyrate producers represent the middle 33% (see table). Each stratification arm will have a minimum of 17 study volunteers bringing the total to n=51. This has been set to ensure the completion of at least 45 volunteers. To optimise equal gender distribution amongst all study arms a minimum of 5 females and 5 males will be recruited for each arm.

Stratification Butyrate range Low ≤13 mM Moderate butyrate 13 - 20mM High butyrate ≥20mM

Primary and secondary outcomes will be analysed between the low and high butyrate producing groups as well as the overall group effect on everyone.

ELIGIBILITY:
Inclusion Criteria:

* i. Men and women aged 18-68 years; BMI ranging from 18-35 kg/m2; measured at the screening visit

Exclusion Criteria:

* i. smokers
* ii. subjects with: diagnosis of diabetes, pregnant, hypertension, renal, hepatic, haematological disease, coronary heart disease or any gastrointestinal disorder
* ii. unsuitable veins for blood sampling;
* iii. inability to speak, read and understand English.
* iv. Use of antibiotics within the last 3 months will automatically exclude volunteers.
* v. Vegans. Fermented whey concentrate, (FWC), is derived from milk (animal product) which excludes potential participants adhering to a vegan diet.
* vi. allergy to any of the following: cow milk, lactose, casein, whey, sucralose, acesulfame K, citric acid, potassium benzoate, fruit flavourings.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2020-04-08 (Actual); Study Completion 2020-04-08 (Actual)

PRIMARY OUTCOMES:
Faecal butyrate concentration - comparing upper and lower tertile of volunteers | Baseline measurement (Visit 1) and end of study (visit 3, 8 weeks later) [Baseline butyrate calculated from the average of two values per individual at Day -7 and Day 0; End of study value is the average from two samples collected at Day 49 and 56
  Change in relative proportion of butyrate (percentage of total SCFA - sum of propionate, butyrate, acetate, valerate, iso-valerate, iso-butyrate, succinate, lactate mM (millimolar values from gas chromatography) and absolute concentration (mM millimolar) when comparing volunteers as stratified by faecal butyrate levels at start of study. A comparison will be made between the butyrate concentration-dependent groupings.
Faecal butyrate concentration - intervention group effect | Baseline measurement (Visit 1) and end of study (visit 3, 8 weeks later) [Baseline butyrate calculated from the average of two values per individual at Day -7 and Day 0; End of study value is the average from two samples collected at Day 49 and 56
  Change in relative proportion of butyrate (percentage of total SCFA) and absolute concentration (mM, millimolar) across the total study group
Microbiota composition change | Assessed as change between day 0 and day 56
  Changes in the composition of the microbiota will be based on next-generation sequence analysis of 16S rRNA (ribosomal ribonucleic acid) genes extracted from faecal samples provided by all volunteers

SECONDARY OUTCOMES:
Gastrointestinal wellness questionnaire | Day 0, 7, 14, 21, 28, 35, 42, 49 and 56
  Changes in frequency or consistency of bowel movements and gastrointestinal well being will be assessed with a self-administered weekly questionnaire (ranked on a linear likert scale).
  The questionnaire asks volunteers to rank nausea, bloating, flatulence, abdominal cramps, rumbling, indigestion, fullness/distension and early satiation over the last 24 hours. The scale is scored from -3 being considerably less, -2 moderately less, -1 for slightly less and 0 for as usual. Responses such as slightly more are scored as 1, moderately more as 2 and considerately more as 3.
  Scores will be aggregated across all categories and compared as a whole to represent general GI wellness changing throughout the intervention.
  Participants have a blank box to fill in with the number of bowel movements in the last 24hr and are asked to rank them on the Bristol stool scale (0-7, visual guide included in the questionnaire). Scores will be assessed as averages over the control and intervention periods.
Glucose tolerance and insulin sensitivity | Measured on Day 0 and Day 56
  Comparison of change in response to Oral glucose tolerance test (3 hours) using the total and incremental area under the curve (AUC)for both glucose and insulin concentrations.
  Both values are measured in arbitrary units and calculated by the standard trapezoid method.
  Incremental AUC is the baseline corrected output for total AUC.
  Comparison will be made between group averages at baseline and post-intervention
Health related quality of life questionnaire | scored on Day 0 and 56
  Change in score in health-related quality of life questionnaire General health is ranked on a scale of excellent, very good, good, fair and poor with scores ranging from 1 - 5 respectively.
  Volunteers are asked to write the relevant days they have been affected by:
  physical health, mental health or impaired by poor mental and physical health, or pain over the last 30 days.
  Participants are asked to respond to the following questions relating to the past 30 days:
  how many days have they felt sad/blue, worried/tense/anxious, did not have enough rest/sleep and have felt very healthy and full of energy.
  Each category will be individually compared at baseline and post-intervention.
Small intestinal fermentation | measured on Days 0, 14 and 56
  Change in Breath test assessment of hydrogen and methane levels (given in ppm - parts per million) and faecal pH (using standard pH meter)
Faecal pH | measured at day 0 and 56
  Change in Faecal pH, using standard pH meter - Scale 0-14
Faecal moisture content | measured at day 0 and 56
  proportion of faeces (in the percentage of total weight) made up of water

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra M Johnstone, PhD, Principal Investigator — University of Aberdeen; Karen P Scott, PhD, Principal Investigator — University of Aberdeen
Locations (1):
- The Rowett Institute, Human Nutrition Unit, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No